CLINICAL TRIAL: NCT03992378
Title: Neuromodulation to Regulate Inflammation and Autonomic Imbalance in Sepsis
Acronym: NERINASEPSIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Oklahoma City VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9227
Record Dates: First submitted 2019-06-05; First posted 2019-06-20 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Septic Shock
Keywords: Sepsis
MeSH Terms: conditions — Shock, Septic; Sepsis

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active Treatment (Experimental): Patients will receive a single 4-hour session of active transcutaneous vagus nerve stimulation.
  Interventions: Device: Low Level Transcutaneous Vagus Nerve Stimulation
- Sham Control (Sham Comparator): Patients will receive a single 4-hour session of sham transcutaneous vagus nerve stimulation.
  Interventions: Device: Low Level Transcutaneous Vagus Nerve Stimulation

INTERVENTIONS:
Device: Low Level Transcutaneous Vagus Nerve Stimulation — Stimulation of the auricular branch of the vagus nerve at tragus of the external ear delivered by Parasym device.
  Arms: Active Treatment
Device: Low Level Transcutaneous Vagus Nerve Stimulation — Stimulation of the ear lobe delivered by Parasym device.
  Arms: Sham Control

SUMMARY:
Sepsis is life-threatening organ dysfunction caused by a dysregulated host response to infection. It is the most expensive healthcare condition to treat in United States and has a mortality rate of nearly 30%. It is widely known that exaggerated inflammation and imbalance between sympathetic and parasympathetic arms of the autonomic nervous system (ANS) contribute to progression and adverse outcomes in sepsis. The role of unchecked inflammation and unregulated ANS as a potential treatment target is an important gap in our knowledge that should be explored.

Cholinergic anti-inflammatory pathway (CAP) is an intricate network where the ANS senses inflammation by vagus nerve afferents and tries to regulate it by vagus nerve efferents to the reticuloendothelial system. The central hypothesis of this pilot clinical trial is that transcutaneous vagus nerve stimulation (TVNS) at tragus of the external ear can activate the CAP to suppress inflammation and improve autonomic imbalance as measured by inflammatory cytokine levels and heart rate variability (HRV) analysis. The investigators plan to randomize patients with septic shock into active and sham stimulation groups and study the effects of vagal stimulation on inflammatory cytokines, HRV and a clinical severity score of sepsis. Both groups will continue to receive the standard of care treatment for sepsis irrespective of group assignments. The investigators hypothesize that 4 hours of TVNS will suppress inflammatory markers and improve the balance between sympathetic and parasympathetic arms of ANS as measured by HRV, resulting in improved Sequential Organ Failure Assessment Score (SOFA). The preliminary data generated from this pilot study will lay the foundation for a larger clinical trial.

ELIGIBILITY:
Inclusion Criteria:

Septic shock (meeting severe sepsis and having persistent systolic blood pressure <90mmHg despite adequate fluid resuscitation).

Exclusion Criteria:

* Unilateral or bilateral vagotomy
* History of myocardial infarction or stroke in the last 1 year
* Recurrent vasovagal syncope
* Sick sinus syndrome without pacemaker
* Bifascicular heart block
* 2nd or 3rd-degree heart block
* Hypotension due to autonomic dysfunction
* Pregnant women
* Prisoners and patients with suicidal ideation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2019-10-10 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Inflammatory Cytokine Tumor Necrosis Factor Alpha | Baseline to 4 hours and baseline to 24 hours post stimulation
  Serum inflammatory cytokine

SECONDARY OUTCOMES:
Change in Heart Rate Variability | Baseline to 4 hours post stimulation
  Time domain and frequency domain measures of heart rate variability
Change in Sequential Organ Failure Assessment Score | Baseline to 24 hours post stimulation
  Sequential Organ Failure Assessment Score calculation

CONTACTS AND LOCATIONS:
Overall Officials: Houssein Youness, MD, Principal Investigator — University of Oklahoma; Zain Ul Abideen Asad, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Derived] Goggins E, Inoue H, Okusa MD. Neuroimmune Control of Inflammation in Acute Kidney Injury and Multiorgan Dysfunction. J Am Soc Nephrol. 2025 Dec 1;36(12):2473-2484. doi: 10.1681/ASN.0000000813. Epub 2025 Jul 7. PMID 40622772